CLINICAL TRIAL: NCT04564209
Title: Information Visualizations to Facilitate Clinician-patient Communication in HIV Care (Info Viz: HIV)
Brief Title: Information Visualizations to Enhance HIV-related Communication
Acronym: Info Viz: HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 20-0163; R00NR017829 (NIH)
Record Dates: First submitted 2020-09-21; First posted 2020-09-25 (Actual); Results first posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: HIV; Communication Research
Keywords: Health literacy; HIV; Infographic; Information-visualization; Clinician-patient communication; Health education
MeSH Terms: conditions — Health Education | interventions — Health

STUDY DESIGN:
Intervention Model Description: There is a treatment and a control group at each site.
Who Masked: Investigator
Masking Description: Study team members who are recruiting will not be aware of which group study participants are being assigned to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): The treatment group will be exposed to the infographic intervention when they present for clinic/study visits. During their visit with the provider, the provider offer health education while using infographics.
  Interventions: Other: Info Viz for Health
- Control (No Intervention): The control groups will receive standard health education.

INTERVENTIONS:
Other: Info Viz for Health — During the intervention, health care providers provide HIV-related health education using a mobile app that contains a bilingual database of relevant infographics.
  Arms: Treatment

SUMMARY:
HIV disproportionately affects Latinos who have more infections, faster disease progression, more HIV-related deaths, and slower diagnosis and treatment than their white/majority counterparts. This is a concern across the United States (US) and in developing countries, such as the Dominican Republic (DR). The HIV-related health disparities experienced by Latinos are made worse when those living with HIV have low health literacy and difficulty understanding the information they need to manage their health.

The PI developed a set of images to assist clinicians in providing information to Latino people living with HIV (PLWH). These images have been put into a mobile health app so clinicians can easily access them during clinic visits. The PI has tested her with PLWH in the DR and in New York City. So, the next steps in this research are to ensure the images are relevant and useful to Latinos across the United States (US) and to further assess if, and to what extent, the images can improve health outcomes among PLWH in the US and in the DR. We will therefore, adapt images to Latinos of Mexican origin/descent and then test them to determine if these images help clinicians provide information to patients by conducting a study at clinical sites in the US and in the DR.

ELIGIBILITY:
Inclusion Criteria:

- Participants must self-identify as Latino, be English or Spanish-speaking, living with HIV with a detectable viral load (>200 copies/mL) at any point in the past year or have an indication of adherence risk, and planning to receive care at the study site for the next year.

Exclusion Criteria:

* Not meeting inclusion criteria or not having the mental capacity to understand the study or provide informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Stonbraker, PhD, MPH, RN, Principal Investigator — University of Colorado College of Nursing
Locations (2):
- Denver Health and Hospital Authority, Denver, Colorado, United States
- Clínica de Familia La Romana, La Romana, Dominican Republic

IPD SHARING:
Plan to Share IPD: Yes
De-identified data of individual participant data will be made available to qualified researchers seeking to replicate methods or to those working on a new study who need the evidence-base to do so in a rigorous way. All de-identified participant data will be shared with other researchers. Please note that much of this data will be in Spanish.
Supporting Information: CSR, Analytic Code
Time Frame: Data will be available 3 months after the publication of primary results.
Access Criteria: To request data please email the study director listed on this record with the reason you need the data and your planned use of it.

REFERENCES:
- [Background] Henao-Martinez AF, Castillo-Mancilla JR. The Hispanic HIV Epidemic. Curr Infect Dis Rep. 2013 Feb;15(1):46-51. doi: 10.1007/s11908-012-0306-0. PMID 23184612
- [Background] Ochoa SC, Sampalis J. Risk perception and vulnerability to STIs and HIV/AIDS among immigrant Latin-American women in Canada. Cult Health Sex. 2014;16(4):412-25. doi: 10.1080/13691058.2014.884632. Epub 2014 Apr 4. PMID 24697557
- [Background] Goldenberg SM, Strathdee SA, Perez-Rosales MD, Sued O. Mobility and HIV in Central America and Mexico: a critical review. J Immigr Minor Health. 2012 Feb;14(1):48-64. doi: 10.1007/s10903-011-9505-2. PMID 21789558
- [Background] Gonzalez JS, Hendriksen ES, Collins EM, Duran RE, Safren SA. Latinos and HIV/AIDS: examining factors related to disparity and identifying opportunities for psychosocial intervention research. AIDS Behav. 2009 Jun;13(3):582-602. doi: 10.1007/s10461-008-9402-4. Epub 2008 May 23. PMID 18498050
- [Background] Xia Q, Braunstein SL, Wiewel EW, Hadler JL, Torian LV. Persistent Racial Disparities in HIV Infection in the USA: HIV Prevalence Matters. J Racial Ethn Health Disparities. 2017 Feb;4(1):87-93. doi: 10.1007/s40615-015-0205-9. Epub 2016 Jan 8. PMID 26746424
- [Background] Rojas P, Malow R, Ruffin B, Rothe EM, Rosenberg R. The HIV/AIDS Epidemic in the Dominican Republic: Key Contributing Factors. J Int Assoc Physicians AIDS Care (Chic). 2011 Sep-Oct;10(5):306-15. doi: 10.1177/1545109710397770. Epub 2011 Mar 2. PMID 21368008
- [Background] De Boni R, Veloso VG, Grinsztejn B. Epidemiology of HIV in Latin America and the Caribbean. Curr Opin HIV AIDS. 2014 Mar;9(2):192-8. doi: 10.1097/COH.0000000000000031. PMID 24356327
- [Background] Perez-Escamilla R. Acculturation, nutrition, and health disparities in Latinos. Am J Clin Nutr. 2011 May;93(5):1163S-7S. doi: 10.3945/ajcn.110.003467. Epub 2011 Mar 2. PMID 21367946
- [Background] Barreto SM, Miranda JJ, Figueroa JP, Schmidt MI, Munoz S, Kuri-Morales PP, Silva JB Jr. Epidemiology in Latin America and the Caribbean: current situation and challenges. Int J Epidemiol. 2012 Apr;41(2):557-71. doi: 10.1093/ije/dys017. Epub 2012 Mar 9. PMID 22407860
- [Background] Wawrzyniak AJ, Ownby RL, McCoy K, Waldrop-Valverde D. Health literacy: impact on the health of HIV-infected individuals. Curr HIV/AIDS Rep. 2013 Dec;10(4):295-304. doi: 10.1007/s11904-013-0178-4. PMID 24222474
- [Background] Laws MB, Lee Y, Rogers WH, Beach MC, Saha S, Korthuis PT, Sharp V, Cohn J, Moore R, Wilson IB. Provider-patient communication about adherence to anti-retroviral regimens differs by patient race and ethnicity. AIDS Behav. 2014 Jul;18(7):1279-87. doi: 10.1007/s10461-014-0697-z. PMID 24464408
- [Background] Kalichman SC, Rompa D. Functional health literacy is associated with health status and health-related knowledge in people living with HIV-AIDS. J Acquir Immune Defic Syndr. 2000 Dec 1;25(4):337-44. doi: 10.1097/00042560-200012010-00007. PMID 11114834
- [Background] Kalichman SC, Benotsch E, Suarez T, Catz S, Miller J, Rompa D. Health literacy and health-related knowledge among persons living with HIV/AIDS. Am J Prev Med. 2000 May;18(4):325-31. doi: 10.1016/s0749-3797(00)00121-5. PMID 10788736
- [Background] Zhang NJ, Terry A, McHorney CA. Impact of health literacy on medication adherence: a systematic review and meta-analysis. Ann Pharmacother. 2014 Jun;48(6):741-51. doi: 10.1177/1060028014526562. Epub 2014 Mar 11. PMID 24619949
- [Background] Barlow J, Wright C, Sheasby J, Turner A, Hainsworth J. Self-management approaches for people with chronic conditions: a review. Patient Educ Couns. 2002 Oct-Nov;48(2):177-87. doi: 10.1016/s0738-3991(02)00032-0. PMID 12401421
- [Background] Mackey LM, Doody C, Werner EL, Fullen B. Self-Management Skills in Chronic Disease Management: What Role Does Health Literacy Have? Med Decis Making. 2016 Aug;36(6):741-59. doi: 10.1177/0272989X16638330. Epub 2016 Apr 6. PMID 27053527
- [Background] Becerra BJ, Arias D, Becerra MB. Low Health Literacy among Immigrant Hispanics. J Racial Ethn Health Disparities. 2017 Jun;4(3):480-483. doi: 10.1007/s40615-016-0249-5. Epub 2016 Jun 20. PMID 27324821
- [Background] Schulman-Green D, Jaser S, Martin F, Alonzo A, Grey M, McCorkle R, Redeker NS, Reynolds N, Whittemore R. Processes of self-management in chronic illness. J Nurs Scholarsh. 2012 Jun;44(2):136-44. doi: 10.1111/j.1547-5069.2012.01444.x. Epub 2012 May 2. PMID 22551013
- [Background] Rao JK, Anderson LA, Inui TS, Frankel RM. Communication interventions make a difference in conversations between physicians and patients: a systematic review of the evidence. Med Care. 2007 Apr;45(4):340-9. doi: 10.1097/01.mlr.0000254516.04961.d5. PMID 17496718
- [Background] Stonbraker S, Smaldone A, Luft H, Cushman LF, Lerebours Nadal L, Halpern M, Larson E. Associations between health literacy, HIV-related knowledge, and information behavior among persons living with HIV in the Dominican Republic. Public Health Nurs. 2018 May;35(3):166-175. doi: 10.1111/phn.12382. Epub 2017 Dec 29. PMID 29285785
- [Background] Stonbraker S, Befus M, Lerebours Nadal L, Halpern M, Larson E. Factors Associated with Health Information Seeking, Processing, and Use Among HIV Positive Adults in the Dominican Republic. AIDS Behav. 2017 Jun;21(6):1588-1600. doi: 10.1007/s10461-016-1569-5. PMID 27714522
- [Background] Stonbraker S, Larson E. Health-information needs of HIV-positive adults in Latin America and the Caribbean: an integrative review of the literature. AIDS Care. 2016 Oct;28(10):1223-9. doi: 10.1080/09540121.2016.1173645. Epub 2016 Apr 21. PMID 27098484
- [Background] Stonbraker S, Halpern M, Bakken S, Schnall R. Developing Infographics to Facilitate HIV-Related Patient-Provider Communication in a Limited-Resource Setting. Appl Clin Inform. 2019 Aug;10(4):597-609. doi: 10.1055/s-0039-1694001. Epub 2019 Aug 14. PMID 31412382
- [Background] Stonbraker S, Richards S, Halpern M, Bakken S, Schnall R. Priority Topics for Health Education to Support HIV Self-Management in Limited-Resource Settings. J Nurs Scholarsh. 2019 Mar;51(2):168-177. doi: 10.1111/jnu.12448. Epub 2018 Nov 19. PMID 30450740
- [Background] Garcia-Retamero R, Okan Y, Cokely ET. Using visual aids to improve communication of risks about health: a review. ScientificWorldJournal. 2012;2012:562637. doi: 10.1100/2012/562637. Epub 2012 May 2. PMID 22629146
- [Background] Garcia-Retamero R, Dhami MK. Pictures speak louder than numbers: on communicating medical risks to immigrants with limited non-native language proficiency. Health Expect. 2011 Mar;14 Suppl 1(Suppl 1):46-57. doi: 10.1111/j.1369-7625.2011.00670.x. PMID 21323820
- [Background] Houts PS, Doak CC, Doak LG, Loscalzo MJ. The role of pictures in improving health communication: a review of research on attention, comprehension, recall, and adherence. Patient Educ Couns. 2006 May;61(2):173-90. doi: 10.1016/j.pec.2005.05.004. Epub 2005 Aug 24. PMID 16122896
- [Background] Arcia A, Suero-Tejeda N, Bales ME, Merrill JA, Yoon S, Woollen J, Bakken S. Sometimes more is more: iterative participatory design of infographics for engagement of community members with varying levels of health literacy. J Am Med Inform Assoc. 2016 Jan;23(1):174-83. doi: 10.1093/jamia/ocv079. Epub 2015 Jul 13. PMID 26174865
- [Background] Kreuter MW, Lukwago SN, Bucholtz RD, Clark EM, Sanders-Thompson V. Achieving cultural appropriateness in health promotion programs: targeted and tailored approaches. Health Educ Behav. 2003 Apr;30(2):133-46. doi: 10.1177/1090198102251021. PMID 12693519
- [Background] Kreuter MW, Strecher VJ, Glassman B. One size does not fit all: the case for tailoring print materials. Ann Behav Med. 1999 Fall;21(4):276-83. doi: 10.1007/BF02895958. PMID 10721433
- [Background] Fernandez-Rhodes L, Robinson WR, Sotres-Alvarez D, Franceschini N, Castaneda SF, Buelna C, Moncrieft A, Llabre M, Daviglus ML, Qi Q, Agarwal A, Isasi CR, Smokowski P, Gordon-Larsen P, North KE. Accuracy of Self-reported Weight in Hispanic/Latino Adults of the Hispanic Community Health Study/Study of Latinos. Epidemiology. 2017 Nov;28(6):847-853. doi: 10.1097/EDE.0000000000000728. PMID 28767517
- [Background] Dillard PK, Zuniga JA, Holstad MM. An integrative review of the efficacy of motivational interviewing in HIV management. Patient Educ Couns. 2017 Apr;100(4):636-646. doi: 10.1016/j.pec.2016.10.029. Epub 2016 Nov 8. PMID 27838113
- [Background] Mandel JC, Kreda DA, Mandl KD, Kohane IS, Ramoni RB. SMART on FHIR: a standards-based, interoperable apps platform for electronic health records. J Am Med Inform Assoc. 2016 Sep;23(5):899-908. doi: 10.1093/jamia/ocv189. Epub 2016 Feb 17. PMID 26911829
- [Background] Sullivan PS, Purcell DW, Grey JA, Bernstein KT, Gift TL, Wimbly TA, Hall E, Rosenberg ES. Patterns of Racial/Ethnic Disparities and Prevalence in HIV and Syphilis Diagnoses Among Men Who Have Sex With Men, 2016: A Novel Data Visualization. Am J Public Health. 2018 Nov;108(S4):S266-S273. doi: 10.2105/AJPH.2018.304762. PMID 30383430
- [Background] Vega WA, Rodriguez MA, Gruskin E. Health disparities in the Latino population. Epidemiol Rev. 2009;31:99-112. doi: 10.1093/epirev/mxp008. Epub 2009 Aug 27. PMID 19713270
- [Background] Osborn CY, Paasche-Orlow MK, Davis TC, Wolf MS. Health literacy: an overlooked factor in understanding HIV health disparities. Am J Prev Med. 2007 Nov;33(5):374-8. doi: 10.1016/j.amepre.2007.07.022. PMID 17950402
- [Background] Berkman ND, Sheridan SL, Donahue KE, Halpern DJ, Crotty K. Low health literacy and health outcomes: an updated systematic review. Ann Intern Med. 2011 Jul 19;155(2):97-107. doi: 10.7326/0003-4819-155-2-201107190-00005. PMID 21768583
- [Background] Iribarren S, Siegel K, Hirshfield S, Olender S, Voss J, Krongold J, Luft H, Schnall R. Self-Management Strategies for Coping with Adverse Symptoms in Persons Living with HIV with HIV Associated Non-AIDS Conditions. AIDS Behav. 2018 Jan;22(1):297-307. doi: 10.1007/s10461-017-1786-6. PMID 28488165
- [Background] Millard T, Elliott J, Girdler S. Self-management education programs for people living with HIV/AIDS: a systematic review. AIDS Patient Care STDS. 2013 Feb;27(2):103-13. doi: 10.1089/apc.2012.0294. Epub 2013 Jan 8. PMID 23298279
- [Background] McMahon T, Ward PR. HIV among immigrants living in high-income countries: a realist review of evidence to guide targeted approaches to behavioural HIV prevention. Syst Rev. 2012 Nov 20;1:56. doi: 10.1186/2046-4053-1-56. PMID 23168134
- [Background] Sauceda JA, Brooks RA, Xavier J, Maiorana A, Georgetti Gomez L, Zamudio-Haas S, Rodriguez-Diaz CE, Cajina A, Myers J. From Theory to Application: A Description of Transnationalism in Culturally-Appropriate HIV Interventions of Outreach, Access, and Retention Among Latino/a Populations. J Immigr Minor Health. 2019 Apr;21(2):332-345. doi: 10.1007/s10903-018-0753-2. PMID 29767401
- [Background] Kasper J, van de Roemer A, Pottgen J, Rahn A, Backhus I, Bay Y, Kopke S, Heesen C. A new graphical format to communicate treatment effects to patients-A web-based randomized controlled trial. Health Expect. 2017 Aug;20(4):797-804. doi: 10.1111/hex.12522. Epub 2016 Dec 16. PMID 27981688
- [Background] Storey D, Seifert-Ahanda K, Andaluz A, Tsoi B, Matsuki JM, Cutler B. What is health communication and how does it affect the HIV/AIDS continuum of care? A brief primer and case study from New York City. J Acquir Immune Defic Syndr. 2014 Aug 15;66 Suppl 3:S241-9. doi: 10.1097/QAI.0000000000000243. PMID 25007193
- [Background] Sorlie V, Lopez RA. When language, health literacy, and miscommunication collide: tremors versus seizures. Fam Med. 2011 Jan;43(1):48-50. No abstract available. PMID 21213140
- [Background] Zolnierek KB, Dimatteo MR. Physician communication and patient adherence to treatment: a meta-analysis. Med Care. 2009 Aug;47(8):826-34. doi: 10.1097/MLR.0b013e31819a5acc. PMID 19584762
- [Background] Mogobe KD, Shaibu S, Matshediso E, Sabone M, Ntsayagae E, Nicholas PK, Portillo CJ, Corless IB, Rose CD, Johnson MO, Webel A, Cuca Y, Rivero-Mendez M, Solis Baez SS, Nokes K, Reyes D, Kemppainen J, Reid P, Sanzero Eller L, Lindgren T, Holzemer WL, Wantland D. Language and Culture in Health Literacy for People Living with HIV: Perspectives of Health Care Providers and Professional Care Team Members. AIDS Res Treat. 2016;2016:5015707. doi: 10.1155/2016/5015707. Epub 2016 Jun 2. PMID 27340564
- [Background] Grodensky CA, Golin CE, Pack AP, Pettifor A, Demers M, Massa C, Kamanga G, McKenna K, Corneli A. Adaptation and delivery of a motivational interviewing-based counseling program for persons acutely infected with HIV in Malawi: Implementation and lessons learned. Patient Educ Couns. 2018 Jun;101(6):1103-1109. doi: 10.1016/j.pec.2018.02.004. Epub 2018 Feb 7. PMID 29519656
- [Background] Beach MC, Laws MB, Rose G, Roter D, Lee Y, Chander G, Woodson T, Moore RD, Rogers W, Wilson IB. Effects of Minimal Versus Intensive Intervention to Enhance Motivational Interviewing in HIV Care. AIDS Behav. 2018 Jan;22(1):276-286. doi: 10.1007/s10461-017-1794-6. PMID 28578544
- [Background] Chang BL, Bakken S, Brown SS, Houston TK, Kreps GL, Kukafka R, Safran C, Stavri PZ. Bridging the digital divide: reaching vulnerable populations. J Am Med Inform Assoc. 2004 Nov-Dec;11(6):448-57. doi: 10.1197/jamia.M1535. Epub 2004 Aug 6. PMID 15299002
- [Background] Levy H, Janke AT, Langa KM. Health literacy and the digital divide among older Americans. J Gen Intern Med. 2015 Mar;30(3):284-9. doi: 10.1007/s11606-014-3069-5. Epub 2014 Nov 12. PMID 25387437
- [Background] Syzdykova A, Malta A, Zolfo M, Diro E, Oliveira JL. Open-Source Electronic Health Record Systems for Low-Resource Settings: Systematic Review. JMIR Med Inform. 2017 Nov 13;5(4):e44. doi: 10.2196/medinform.8131. PMID 29133283
- [Background] Wilson BD, Miller RL. Examining strategies for culturally grounded HIV prevention: a review. AIDS Educ Prev. 2003 Apr;15(2):184-202. doi: 10.1521/aeap.15.3.184.23838. PMID 12739794
- [Background] Lescano CM, Brown LK, Raffaelli M, Lima LA. Cultural factors and family-based HIV prevention intervention for Latino youth. J Pediatr Psychol. 2009 Nov-Dec;34(10):1041-52. doi: 10.1093/jpepsy/jsn146. Epub 2009 Jan 30. PMID 19181820
- [Background] Devieux JG, Malow RM, Jean-Gilles MM, Samuels DM, Deschamps MM, Ascencio M Jr, Jean-Baptiste L, Pape JW. Reducing health disparities through culturally sensitive treatment for HIV+ adults in Haiti. ABNF J. 2004 Nov-Dec;15(6):109-15. PMID 18399360
- [Background] Ramos Z, Alegria M. Cultural adaptation and health literacy refinement of a brief depression intervention for Latinos in a low-resource setting. Cultur Divers Ethnic Minor Psychol. 2014 Apr;20(2):293-301. doi: 10.1037/a0035021. Epub 2014 Mar 3. PMID 24588455
- [Background] Sarkar U, Gourley GI, Lyles CR, Tieu L, Clarity C, Newmark L, Singh K, Bates DW. Usability of Commercially Available Mobile Applications for Diverse Patients. J Gen Intern Med. 2016 Dec;31(12):1417-1426. doi: 10.1007/s11606-016-3771-6. Epub 2016 Jul 14. PMID 27418347
- [Background] Abraido-Lanza AF, Echeverria SE, Florez KR. Latino Immigrants, Acculturation, and Health: Promising New Directions in Research. Annu Rev Public Health. 2016;37:219-36. doi: 10.1146/annurev-publhealth-032315-021545. Epub 2016 Jan 6. PMID 26735431
- [Background] Eisinger RW, Dieffenbach CW, Fauci AS. HIV Viral Load and Transmissibility of HIV Infection: Undetectable Equals Untransmittable. JAMA. 2019 Feb 5;321(5):451-452. doi: 10.1001/jama.2018.21167. No abstract available. PMID 30629090
- [Background] Gearing RE, El-Bassel N, Ghesquiere A, Baldwin S, Gillies J, Ngeow E. Major ingredients of fidelity: a review and scientific guide to improving quality of intervention research implementation. Clin Psychol Rev. 2011 Feb;31(1):79-88. doi: 10.1016/j.cpr.2010.09.007. Epub 2010 Oct 7. PMID 21130938
- [Background] Toren KG, Buskin SE, Dombrowski JC, Cassels SL, Golden MR. Time From HIV Diagnosis to Viral Load Suppression: 2007-2013. Sex Transm Dis. 2016 Jan;43(1):34-40. doi: 10.1097/OLQ.0000000000000376. PMID 26650994
- [Background] Street RL Jr, Makoul G, Arora NK, Epstein RM. How does communication heal? Pathways linking clinician-patient communication to health outcomes. Patient Educ Couns. 2009 Mar;74(3):295-301. doi: 10.1016/j.pec.2008.11.015. Epub 2009 Jan 15. PMID 19150199
- [Background] Lee SY, Stucky BD, Lee JY, Rozier RG, Bender DE. Short Assessment of Health Literacy-Spanish and English: a comparable test of health literacy for Spanish and English speakers. Health Serv Res. 2010 Aug;45(4):1105-20. doi: 10.1111/j.1475-6773.2010.01119.x. Epub 2010 May 24. PMID 20500222
- [Background] Weiss BD, Mays MZ, Martz W, Castro KM, DeWalt DA, Pignone MP, Mockbee J, Hale FA. Quick assessment of literacy in primary care: the newest vital sign. Ann Fam Med. 2005 Nov-Dec;3(6):514-22. doi: 10.1370/afm.405. PMID 16338915
- [Background] Chen WT, Wantland D, Reid P, Corless IB, Eller LS, Iipinge S, Holzemer WL, Nokes K, Sefcik E, Rivero-Mendez M, Voss J, Nicholas P, Phillips JC, Brion JM, Rose CD, Portillo CJ, Kirksey K, Sullivan KM, Johnson MO, Tyer-Viola L, Webel AR. Engagement with Health Care Providers Affects Self- Efficacy, Self-Esteem, Medication Adherence and Quality of Life in People Living with HIV. J AIDS Clin Res. 2013 Nov 1;4(11):256. doi: 10.4172/2155-6113.1000256. PMID 24575329
- [Background] Ritter PL, Lorig K. The English and Spanish Self-Efficacy to Manage Chronic Disease Scale measures were validated using multiple studies. J Clin Epidemiol. 2014 Nov;67(11):1265-73. doi: 10.1016/j.jclinepi.2014.06.009. Epub 2014 Aug 3. PMID 25091546
- [Background] Knobel H, Alonso J, Casado JL, Collazos J, Gonzalez J, Ruiz I, Kindelan JM, Carmona A, Juega J, Ocampo A; GEEMA Study Group. Validation of a simplified medication adherence questionnaire in a large cohort of HIV-infected patients: the GEEMA Study. AIDS. 2002 Mar 8;16(4):605-13. doi: 10.1097/00002030-200203080-00012. PMID 11873004
- [Background] Monroe AK, Pena JS, Moore RD, Riekert KA, Eakin MN, Kripalani S, Chander G. Randomized controlled trial of a pictorial aid intervention for medication adherence among HIV-positive patients with comorbid diabetes or hypertension. AIDS Care. 2018 Feb;30(2):199-206. doi: 10.1080/09540121.2017.1360993. Epub 2017 Aug 10. PMID 28793785
- [Background] Penn AW, Azman H, Horvath H, Taylor KD, Hickey MD, Rajan J, Negussie EK, Doherty M, Rutherford GW. Supportive interventions to improve retention on ART in people with HIV in low- and middle-income countries: A systematic review. PLoS One. 2018 Dec 14;13(12):e0208814. doi: 10.1371/journal.pone.0208814. eCollection 2018. PMID 30550574

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment | Control
Started | 83 | 81
Completed | 65 | 69
Not Completed | 18 | 12

BASELINE CHARACTERISTICS:
Population: Patient participants for the RCT were adult (≥ 18 years), Hispanic/Latino, English or Spanish-speaking, living with HIV with a detectable viral load (>30 or >40 copies/mL depending on the laboratory test) at any point in the past year or be newly diagnosed with HIV, or have an indication of adherence risk as identified by their provider and be planning to receive care at the study site for the next year. If patient participants are pregnant, they may still be included in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 83 | 81 | 164
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 81 | 79 | 160
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.98 (12.55) | 40.53 (11.10) | 41.77 (11.88)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 23 | 20 | 43
  Female | 60 | 60 | 120
  Other | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 83 | 81 | 164
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 25 | 46
  White | 22 | 15 | 37
  More than one race | 26 | 26 | 52
  Unknown or Not Reported | 14 | 15 | 29
Region of Enrollment [Number; unit: participants]
  United States | 42 | 40 | 82
  Dominican Republic | 41 | 41 | 82
Health Literacy [Count of Participants; unit: Participants] — Health literacy at baseline was assessed with the Short Assessment of Health Literacy - Spanish and English. The number reported is the number of treatment and control participants who scored >= 15 points on this assessment and are considered "likely to be health literate"
  Participants | 47 | 47 | 94

OUTCOME MEASURES:

1. Primary Outcome: Change in CD4 Count Over Time
Description: Change in Cluster of Differentiation 4 (CD4) count measured at 3-month intervals following baseline visit
Time Frame: Baseline, 3-month, 6-month, 9-month
Population: There was some attrition over time.
Measure: Mean (Standard Deviation); unit: Cells/mm3
Arm/Group | Treatment | Control
Number analyzed (Participants) | 83 | 81
Cells/mm3
  Baseline | 446.71 (291.298) | 453.99 (319.543)
  3-Month: number analyzed (Participants) | 79 | 77
  3-Month | 498.04 (313.080) | 537.90 (855.711)
  6-Month: number analyzed (Participants) | 75 | 73
  6-Month | 517.77 (301.422) | 449.14 (263.617)
  9-Month: number analyzed (Participants) | 65 | 69
  9-Month | 505.05 (295.086) | 461.71 (281.784)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority; p = .455, ANOVA

2. Secondary Outcome: Change in Viral Load Over Time
Description: Change in viral load count measured at 3-month intervals following baseline
Time Frame: Baseline, 3-month, 6-month, 9-month
Population: There was some attrition over time.
Measure: Mean (Standard Deviation); unit: copies/mL
Arm/Group | Treatment | Control
Number analyzed (Participants) | 83 | 81
copies/mL
  Baseline | 78824.11 (236642.836) | 63904.54 (234399.365)
  3 Month: number analyzed (Participants) | 79 | 77
  3 Month | 12522.70 (50299.069) | 30596.87 (110589.762)
  6 Month: number analyzed (Participants) | 75 | 74
  6 Month | 4369.15 (17184.787) | 26125.96 (117233.253)
  9 Month: number analyzed (Participants) | 65 | 69
  9 Month | 6057.83 (39523.642) | 19439.14 (96963.360)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority; p = .415, ANOVA

3. Secondary Outcome: HIV-related Knowledge Assessment
Description: 14 questions pertaining to HIV-related knowledge were developed according to the information that will be included in the intervention. Participants will receive one point for each correct answer and then the scores for each question will be summed to obtain a final score. Therefore, the minimum score will be 0 and maximum score will be 14 where the scores closer to 14 indicate patients have more HIV-related knowledge
Time Frame: Baseline, 3-month, 6-month, 9-month
Population: There was some attrition over time.
Measure: Mean (Standard Deviation); unit: HIV-related Knowledge Assessment Scores
Arm/Group | Treatment | Control
Number analyzed (Participants) | 83 | 81
HIV-related Knowledge Assessment Scores
  Baseline | 10.0843 (1.97672) | 10.8210 (2.05595)
  3 Month: number analyzed (Participants) | 79 | 77
  3 Month | 11.7975 (1.59831) | 11.4091 (1.80592)
  6 Month: number analyzed (Participants) | 75 | 74
  6 Month | 12.1867 (1.39684) | 11.7230 (1.62629)
  9 Month: number analyzed (Participants) | 65 | 69
  9 Month | 12.2692 (1.72997) | 12.0435 (1.55000)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority; p = .443, ANOVA

4. Secondary Outcome: Satisfaction With Provider Scale Score
Description: Satisfaction with provider was measured with the Overall Satisfaction with Provider and Clinic scale published by Dang et al., 2016. We asked a selection of questions from this scale based on their appropriateness for our study. The questions asked and the range of possible scores are as follows.
  Question 1: 1 - 7 Question 2: 1 - 10 Question 3: 1 - 7 Question 4: 1 - 5
  Total scores are then calculated by adding participant responses on each of the four questions. The total possible score range for the questions asked from this scale was 4 - 29, with higher scores indicating more satisfaction with HIV provider.
Time Frame: Baseline, 3-month, 6-month, 9-month
Population: There was some attrition over time.
Measure: Mean (Standard Deviation); unit: Satisfaction with provider scale score
Arm/Group | Treatment | Control
Number analyzed (Participants) | 83 | 81
Satisfaction with provider scale score
  Baseline | 27.5783 (2.36911) | 27.4877 (2.61483)
  3 Month: number analyzed (Participants) | 79 | 77
  3 Month | 28.4430 (0.82814) | 27.8961 (2.02994)
  6 Month: number analyzed (Participants) | 75 | 74
  6 Month | 28.2933 (1.45911) | 28.0405 (1.80136)
  9 Month: number analyzed (Participants) | 65 | 69
  9 Month | 28.4923 (1.37071) | 28.1884 (1.81720)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority; p = .457, ANOVA

5. Secondary Outcome: SEMCD Scale Score
Description: The Self#Efficacy for Managing Chronic Disease (SEMCD) scale is a 6#item questionnaire that measures confidence in one's ability to manage fatigue, pain, emotional distress, and other symptoms using self#management techniques.
  Each item is scored from a minimum value of 1 which indicates "not at all confident" to a maximum score of 10, which indicates "completely confident." Final scores are calculated as the mean of the 6 questions ranging from 1(minimum) to 10 (maximum), where higher scores indicate higher self-efficacy (better outcome).
Time Frame: Baseline, 3-month, 6-month, 9-month
Population: There was some attrition over time.
Measure: Mean (Standard Deviation); unit: SEMCD Scale Score
Arm/Group | Treatment | Control
Number analyzed (Participants) | 83 | 81
SEMCD Scale Score
  Baseline: number analyzed (Participants) | 82 | 81
  Baseline | 8.6174 (1.52319) | 8.4372 (1.53408)
  3 Month: number analyzed (Participants) | 79 | 77
  3 Month | 9.0011 (1.30174) | 8.6147 (1.63579)
  6 Month: number analyzed (Participants) | 75 | 73
  6 Month | 9.1678 (1.05592) | 8.8276 (1.25087)
  9 Month: number analyzed (Participants) | 65 | 69
  9 Month | 9.0141 (1.18215) | 8.6860 (1.55831)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority; p = .099, ANOVA

6. Secondary Outcome: Simplified Medication Adherence Questionnaire (SMAQ)
Description: We measured adherence to prescribed antiretroviral therapy with the validated simplified medication adherence questionnaire (SMAQ) (Knobel 2002). This is a 6- item questionnaire that measures medication adherence. There is no minimum or maximum score on this scale. Participants are considered either "adherent" (better outcome) or "non-adherent" (worse outcome) based on their responses to these 6 questions.
  They are considered "non-adherent" if they answer "yes" to questions 1, 2, 3, OR 5, regardless of their answers on the other questions.
  Participants are also considered "non-adherent" when they indicate that they have missed more than two doses of their medication in the past week (response to question 4), or over 2 days of total non-medication during the past 3 months (response on question 6).
Time Frame: Baseline, 3-month, 6-month, 9-month
Population: There was some attrition over time.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control
Number analyzed (Participants) | 83 | 81
Participants
  Baseline: Adherent | 35 | 30
  Baseline: Non Adherent | 48 | 51
  3 Month: number analyzed (Participants) | 79 | 77
  3 Month: Adherent | 35 | 35
  3 Month: Non Adherent | 44 | 42
  6 Month: number analyzed (Participants) | 75 | 74
  6 Month: Adherent | 48 | 37
  6 Month: Non Adherent | 27 | 37
  9 Month: number analyzed (Participants) | 65 | 69
  9 Month: Adherent | 29 | 32
  9 Month: Non Adherent | 36 | 37
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority; p = .338, ANOVA

7. Secondary Outcome: Health Status Average Score
Description: Health status will be assessed with a question on the health status assessment scale, on which participants rank their current health status on a scale of 0 - 100 where 0=death or worst possible health and 100=perfect or best possible health (without HIV infection).
Time Frame: Baseline, 3-month, 6-month, 9-month
Population: There was some attrition over time.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 83 | 81
score on a scale
  Baseline | 84.34 (17.950) | 85.33 (14.374)
  3 Month: number analyzed (Participants) | 79 | 77
  3 Month | 89.52 (13.292) | 87.09 (17.853)
  6 Month: number analyzed (Participants) | 75 | 74
  6 Month | 92.47 (11.129) | 92.38 (11.225)
  9 Month: number analyzed (Participants) | 65 | 69
  9 Month | 91.52 (14.664) | 90.67 (14.060)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority; p = .723, ANOVA

8. Secondary Outcome: Satisfaction With Clinic
Description: Satisfaction with clinic was measured with a selection of questions from the Overall Satisfaction with Provider and Clinic scale published by Dang et al., 2016. To assess satisfaction with the clinics, we asked a selection of questions from this scale based on their appropriateness for our study. The included questions and the associated range of possible scores are as follows.
  Question 7: 1 - 7 points possible Question 8: 1 - 7 points possible Question 9: 1 - 5 points possible
  Total scores are then calculated by adding participant responses on each of the three questions. The total possible score range for the questions asked from this scale was 3 - 19, with higher scores indicating more satisfaction with the clinic.
Time Frame: Baseline, 3-, 6-, and 9-months
Population: There was some attrition over time.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 83 | 81
score on a scale
  Baseline | 18.1 (1.4) | 18.2 (1.1)
  3-months: number analyzed (Participants) | 79 | 77
  3-months | 18.7 (0.6) | 18.5 (1.0)
  6-months: number analyzed (Participants) | 75 | 74
  6-months | 18.7 (0.7) | 18.6 (1.0)
  9-months: number analyzed (Participants) | 65 | 69
  9-months | 18.6 (1.0) | 18.5 (1.0)

9. Other Pre Specified Outcome: Health Literacy Score: Short Assessment of Health Literacy Spanish & English (SAHL S&E)
Description: Health literacy will be assessed using the short assessment of health literacy- Spanish. Scores range from 0 - 18 and a score above a 15 indicates that participants are likely to have adequate health literacy.
Time Frame: Baseline visit only
Measure: Mean (Standard Deviation); unit: Health Literacy Score
Arm/Group | Treatment | Control
Number analyzed (Participants) | 83 | 81
Health Literacy Score | 12.41 (6.280) | 12.81 (6.062)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority; p = .578, t-test, 2 sided

10. Other Pre Specified Outcome: Health Literacy Score: Newest Vital Sign (NVS)
Description: A second measure of health literacy, the Newest Vital Sign (NVS) will also be administered. Scores on this scale range from 0-6 where a score of 0-1 suggests high likelihood of limited literacy, a score of 2-3 indicates the possibility of limited literacy, and a score of 4-6 almost always indicates adequate literacy.
Time Frame: Baseline visit only
Measure: Mean (Standard Deviation); unit: Health Literacy Score: Newest Vital Sign
Arm/Group | Treatment | Control
Number analyzed (Participants) | 83 | 81
Health Literacy Score: Newest Vital Sign | 1.37 (1.998) | 1.41 (2.017)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority; p = .998, t-test, 2 sided

11. Other Pre Specified Outcome: Brief Acculturation Rating Scale for Mexican Americans-II
Description: The Brief Acculturation Rating Scale for Mexican Americans- II (ARMSA-II) is a 12-item scale that measures acculturation with 6 items from the AOS (Anglo Oriented Scale) of the ARSMA-II and 6 items from the MOS (Mexican Oriented Scale) (Bauman 2005). Responses are collected with Likert-type questions on which the scores range from 1 (not at all) to 5 (almost always/extremely often) on each item. The ARMSA-II has been used in Mexican Americans as well as other Latino subgroups, including Dominicans.
  Scores are calculated by summing the scores on each of the six item subscales and then dividing by 12 to get a mean acculturation score. Therefore, the possible range of scores is 1-5 with higher scores indicating greater acculturation.
  Note: The scale was only administered to participants who were not born in the country where data collection took place.
Time Frame: Baseline visit only
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control
Number analyzed (Participants) | 42 | 40
score on a scale | 2.64 (1.48) | 2.70 (1.52)
Statistical Analysis 1: Comparison: Treatment vs Control; Test type: Superiority; p = .864, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Full duration of enrollment (approx 9-18 months).
Description: We used the same definitions as clinicaltrials.gov for adverse event reporting.
Arm/Group | Treatment | Control
All-Cause Mortality (participants affected / at risk) | 1/83 | 1/81
Serious Adverse Events (participants affected / at risk) | 0/83 | 0/81
Other Adverse Events (participants affected / at risk) | 0/83 | 0/81

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-20): https://cdn.clinicaltrials.gov/large-docs/09/NCT04564209/Prot_SAP_001.pdf
  • Informed Consent Form (2022-01-04): https://cdn.clinicaltrials.gov/large-docs/09/NCT04564209/ICF_000.pdf